CLINICAL TRIAL: NCT06000527
Title: Juvenile Recurrent Respiratory Papillomatosis: Establishment of a French National Cohort (PRR : National Cohort " REPA ")
Acronym: REPA
Status: Recruiting | Type: Observational
Sponsor: Imagine Institute (Other)
Responsible Party: Sponsor
Other Study IDs: HJ-20-REPA
Record Dates: First submitted 2023-08-04; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Juvenile Recurrent Respiratory Papillomatosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Recurrent respiratory papillomatosis (RRP) is a rare disease. However, it is the most common benign laryngeal tumor in children. To date, no epidemiological data are available in France. The aim of this study is to establish the epidemiology of juvenile PPR.

DETAILED DESCRIPTION:
Recurrent respiratory papillomatosis (RRP) is characterized by the recurrent proliferation of multiple polypoid squamous tumors in the respiratory tract, linked to HPV infection. RRP is a rare disease. However, it is the most common benign laryngeal tumor in children.

There are currently no French national epidemiological data on this disease. The data collected by the reference centers will enable us to gain a better understanding of this pathology in terms of epidemiology, risk factors, genetic susceptibility and clinical manifestations, as well as to significantly study the efficacy of the various existing therapies and preventive measures, in order to establish a clear, standardized and optimal guideline.

ELIGIBILITY:
Inclusion Criteria:

* Patients with juvenile PRR (disease onset before age 18)
* Followed in the :

  * The MALO CRMR
  * One of the MALO network's CCMRs
  * One of the main correspondent centers

Exclusion Criteria:

* Patients objecting to the collection of their personal data
* Parents of minor patients objecting to the collection of their child's personal data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with juvenile PRR in France
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2032-09-30 (Estimated); Study Completion 2032-09-30 (Estimated)

PRIMARY OUTCOMES:
Epidemiology of juvenile RRP in France by clinical information | 10 years
  age at onset of disease, symptoms, severity score, intensity of disease characterized by need for endoscopies
Epidemiology of juvenile PRR in France according to vaccine and adjuvant therapeutic information | 10 years
  Vaccination and adjuvant therapy information
Epidemiology of juvenile PRR in France by paraclinical information | 10 years
  results of pulmonary imaging, genetic, anatomopathological and immunological tests

SECONDARY OUTCOMES:
Define standardized management of juvenile RRP | 10 years
  Correlations between disease progression and frequency of follow-up, as well as treatments implemented (therapeutic or surgical interventions)
Therapeutic management of RRP | 10 years
  * Frequency of therapeutic surgery
  * Use of adjuvant therapies
Prevention of RRP | 10 years
  Analysis of national vaccination coverage with a vaccine immunizing against HPV 6 and 11

CONTACTS AND LOCATIONS:
Locations (1):
- hôpital Necker Enfants malades, Paris, France